CLINICAL TRIAL: NCT01688336
Title: Phase II Single Arm Clinical Trial of FOLFIRINOX for Unresectable Locally Advanced and Borderline Resectable Pancreatic Cancer
Brief Title: FOLFIRINOX for Unresectable Locally Advanced and Borderline Resectable Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Results unlikely to impact treatment patterns. Time to complete not justified.
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LCCC 1105
Record Dates: First submitted 2012-09-14; First posted 2012-09-19 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-10-06 (Actual); Status verified 2017-09

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic; Phase II; FOLFIRINOX; Unresectable; Regimen; First-line; Resectable; Borderline; Oxaliplatin; Leucovorin; Irinotecan; 5FU; Lineberger; University of North Carolina
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — folfirinox; Oxaliplatin; Leucovorin; Irinotecan; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- FOLFIRINOX (Experimental): FOLFIRINOX given to all subjects
  Interventions: Drug: FOLFIRINOX

INTERVENTIONS:
Drug: FOLFIRINOX — FOLFIRINOX will be given intravenously on Days 1, 15, and 28 of each 28 day cycle. Drugs are given in combination in this order:
  * Oxaliplatin (85 mg/m2)
  * Leucovorin (400mg/ m2)
  * Irinotecan (180 mg/m2)
  * 5FU (400mg/m2)bolus then 2400 mg/m2 over 46 hours
  Other Names: FOLFIRINOX is a chemotherapy regimen comprised of the following drugs, given in combination; -Oxaliplatin; -Leucovorin; -Irinotecan; -5FU

SUMMARY:
This single arm, multi-center phase II clinical trial will assess the safety and efficacy of FOLFIRINOX in the first-line setting in patients with unresectable locally advanced (ULA) and borderline resectable (BR) pancreatic cancer.

DETAILED DESCRIPTION:
FOLFIRINOX regimen was recently presented at an international oncology meeting and represents a new standard in the treatment of metastatic pancreatic cancer for selected patients. With improved overall survival (OS) and response rates (RR) in the metastatic setting, we hypothesize that in patients with less tumor burden, this regimen will be safe and well tolerated, improve OS, progression free survival (PFS), and RR, and improve resectability rates, as compared to historical data from standard single agent gemcitabine therapy for unresectable locally advanced (ULA) patients and standard radiation with concurrent 5 fluorouracil (5FU) chemotherapy for borderline resectable (BR) patients. While both ULA and BR patients will be eligible for the present study, our primary objective concerns ULA patients, and we plan to enroll 45 patients in this group.

Patients meeting eligibility criteria will be consented and treated with FOLFIRINOX every 2 weeks (1 cycle = 4 weeks = 2 treatments). Patients will undergo repeat imaging (CT or MRI) every 2 cycles and reassessed for resectability of the tumor. All patients that are not able to undergo surgical resection, due to insufficient down-staging or patient preference, will continue on protocol-based therapy until disease progression, unacceptable toxicity, study withdrawal, or death.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed adenocarcinoma of the pancreas.
* Measurable or non-measurable but evaluable (as determined by Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1]) unresectable locally advanced (ULA) or borderline resectable (BR) disease that is not amenable to curative intent therapy. Baseline CT abdomen and chest (or MRI abdomen) within 28 days prior to initiation of FOLFIRINOX is required.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* No prior chemotherapy or chemoradiotherapy for pancreatic cancer.
* Age ≥ 18 years of age.
* Laboratory requirements at study entry:

  * Hemoglobin ≥ 10 g/dL (transfusions are acceptable)
  * absolute neutrophil count (ANC) ≥ 1.5 x 109/L
  * Platelets ≥ 100 x 109/L
  * Creatinine ≤ 1.5 x upper limit of normal (ULN), or creatinine clearance ≥ 50 mL/min (estimated by Cockcroft-Gault or measured)
  * Total bilirubin ≤ 1.5 x ULN
  * aspartate aminotransferase/Alanine Aminotransferase (AST/ALT) ≤ 3 x ULN
  * Gamma-Glutamyl Transferase (GGT) ≤ 5 x ULN
* Life expectancy of at least 6 months.
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test performed within 14 days prior to initiation of FOLFIRINOX.
* WOCBP and men must agree to use adequate contraception prior to study entry, for the duration of study participation, and 8 weeks after the end of treatment.
* Before patient registration, written informed consent must be given.

Exclusion Criteria:

* Local recurrence or resectable recurrence of pancreatic cancer.
* Other malignancies within the past 3 years except for adequately treated cervical or vulvar carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated >3 years prior to entry is permitted.
* Hypersensitivity to 5FU, oxaliplatin or other platinum agent, or irinotecan or to their excipients. Known dihydropyrimidine dehydrogenase (DPD) enzyme deficiency.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment. Patients are not permitted to participate in another investigational drug study while being treated on this protocol.
* Cardiac disease: Congestive heart failure symptoms > class II New York Heart Association (NYHA). Unstable angina (anginal symptoms at rest) or new onset angina beginning within the last 3 months. Myocardial infarction within the past 6 months. Cardiac ventricular arrhythmias requiring anti-arrhythmic therapy.
* History of or suspected Gilbert's Disease (baseline testing not required).
* Baseline peripheral neuropathy/paresthesia grade ≥ 1.
* Active hepatitis B, unless patient has been on stable meds for at least 2 months (baseline testing not required).
* Active clinically serious infections (> grade 2).
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within the 12 weeks prior to the first dose FOLFIRINOX.
* Evidence or history of bleeding diathesis or coagulopathy. Note: If therapeutic anticoagulation required, the investigator is encouraged to switch patient to (or maintain on) low molecular weight heparin during the trial.
* Major surgery, open biopsy or significant traumatic injury within 8 weeks of first study drug. A core pancreatic or liver biopsy does not preclude the patient from the study.
* Unable or unwilling to discontinue use of ketoconazole or St John's wort. Use of CYP3A4 enzyme-inducing drugs and strong CYP3A4 inhibitors is discouraged, but not contraindicated.
* Active drug or alcohol abuse.
* Pregnant or lactating women.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08-22 (Actual); Study Completion 2016-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Autumn J McRee, MD, Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: UNC Lineberger Comprehensive Cancer Center homepage — http://unclineberger.org/
- See also: National Cancer Institute (NCI) homepage — http://www.cancer.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 11 patients were consented. One patient was consented but not treated due to metastatic disease and one patient was consented and not treated due to disease progression prior to protocol therapy. 9 patients went on study.
Groups:
- FOLFIRINOX: FOLFIRINOX given to all subjects
  FOLFIRINOX: FOLFIRINOX will be given intravenously on Days 1, 15, and 28 of each 28 day cycle. Drugs are given in combination in this order:
  * Oxaliplatin (85 mg/m2)
  * Leucovorin (400mg/ m2)
  * Irinotecan (180 mg/m2)
  * Fluorouracil (5FU) (400mg/m2)bolus then 2400 mg/m2 over 46 hours
Period: Overall Study
Arm/Group | FOLFIRINOX
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- FOLFIRINOX: FOLFIRINOX given to all subjects
  FOLFIRINOX: FOLFIRINOX will be given intravenously on Days 1, 15, and 28 of each 28 day cycle. Drugs are given in combination in this order:
  * Oxaliplatin (85 mg/m2)
  * Leucovorin (400mg/ m2)
  * Irinotecan (180 mg/m2)
  * 5FU (400mg/m2)bolus then 2400 mg/m2 over 46 hours
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 9
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [51 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Median Overall Survival (OS) of FOLFIRINOX in Patients With Unresectable Locally Advanced (ULA) Pancreatic Cancer
Description: All patients who receive at least Day 1 of FOLFIRINOX treatment will be evaluable and followed up for up to 3 years for the primary outcome of overall survival (OS).
Time Frame: Up to 3 years
Population: Patients with unresectable locally advanced pancreatic cancer.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 5
months | 28.5 [6.2 to NA] — Insufficient number of participants with events

2. Secondary Outcome: Overall Survival for Borderline Resectable Patients
Description: All patients who receive at least Day 1 of FOLFIRINOX treatment will be evaluable and followed up for up to 3 years for the outcome of overall survival (OS)
Time Frame: Up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 4
Months | 9.0 [5.8 to 16.2]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Progression free survival will be measured from D1 of treatment until evidence of tumor progression (including clinical deterioration related to the underlying pancreatic cancer, as assessed by the investigator) or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. Patients that are lost to follow-up will be censored
Time Frame: the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 9
Months | 10.7 [2.0 to 24.8]

4. Secondary Outcome: Objective Response Rate
Description: All patients who have received at least one cycle of treatment will be evaluated. Disease will be evaluated per Response Evaluation Criteria in Solid Tumors (RECIST, version 1.1) for target lesions and assessed by CT and/or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  Patients who drop out of the study prior to disease evaluation will not be evaluable for response unless the patient undergoes radiologic evaluation or their disease progresses clinically.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 9
percentage of patients | 11 [0 to 48]

5. Secondary Outcome: Disease Control Rate (DCR)
Description: Disease control rate will be measured by the percentage of patients with responses (CR) and partial responses (PR) and stable disease (SD), per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI and/or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for a Partial Response nor sufficient increase to qualify for Progression of Disease (POD); Complete Response (CR), Disappearance of all target lesions.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 9
percentage of patients | 89 [52 to 100]

6. Secondary Outcome: Rate of Resectability (RR)
Description: Rate of resectability will be evaluated by determining the percentage of patients who were initially deemed to have ULA or borderline resectable (BR) disease and, following any period of treatment, were subsequently deemed to have resectable disease and undergo surgical resection. The denominator will reflect all patients with ULA or BR disease.
Time Frame: Up to 3 years
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 9
percentage of patients | 22 [0 to 60]

7. Other Pre Specified Outcome: Correlation of Tumor Markers (Ca19-9, CEA) With Outcomes (RR, DCR, PFS, and OS).
Description: Tumor markers (Ca19-9, CEA) will be measured at baseline, every eight weeks and at end of treatment, and will be correlated with outcomes resectability response (RR),disease control rate (DCR), progression free survival (PFS) and overall survival (OS).
Time Frame: Up to 3 years
Population: Data were not collected
Arm/Group | FOLFIRINOX
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | FOLFIRINOX
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRINOX (N=9)
Death (General disorders) | 1 — Sudden death not otherwise specified (NOS)
Urinary Tract Infection (Infections and infestations) | 1
Renal Calculi (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRINOX (N=9)
Abdominal Pain (Gastrointestinal disorders) | 3
Alanine Aminotransferase Increased (Investigations) | 3
Alkaline Phosphatase Increased (Investigations) | 6
Anemia (Blood and lymphatic system disorders) | 7
Anorexia (Gastrointestinal disorders) | 1
Aspartate Aminotransferase Increased (Investigations) | 3
Blood Bilirubin Increased (Investigations) | 1
Chills (General disorders) | 1
Creatinine Increased (Investigations) | 2
Diarrhea (Gastrointestinal disorders) | 4
Dysgeusia (Nervous system disorders) | 1
Edema Limbs (General disorders) | 1
Fatigue (General disorders) | 4
Fever (General disorders) | 1
Ggt Increased (Investigations) | 5
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5
Hyperuricemia (Metabolism and nutrition disorders) | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 6
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Insomnia (Psychiatric disorders) | 1
Lipase Increased (Investigations) | 1
Lymphocyte Count Decreased (Investigations) | 2
Mucositis Oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Neutrophil Count Decreased (Investigations) | 8
Peripheral Sensory Neuropathy (Nervous system disorders) | 4
Platelet Count Decreased (Investigations) | 6
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Syncope (Nervous system disorders) | 1
Vaginal Infection (Infections and infestations) | 1
Vomiting (Gastrointestinal disorders) | 1
White Blood Cell Decreased (Investigations) | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes